CLINICAL TRIAL: NCT04075175
Title: A Phase 1 Study in Healthy Subjects to Evaluate the Safety and Pharmacokinetics of a Human Monoclonal Antibody (mAb) S315 Against Diphtheria Toxin
Brief Title: Evaluate the Safety Pharmacokinetics of a Human Monoclonal Antibody S315 Against Diphtheria Toxin in Healthy Subjects
Acronym: S315
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MassBiologics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: MBL-DIPH-19-01
Record Dates: First submitted 2019-08-15; First posted 2019-08-30 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Diphtheria
MeSH Terms: conditions — Diphtheria | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S315 human monoclonal antibody (Experimental): 5 cohorts of 8 subjects each randomized 6:2 (S315:Placebo (0.9% Sodium Chloride)) with escalation of a fixed dose of S315
  Interventions: Drug: S315
- 0.9% sodium chloride (NaCl) (Placebo Comparator): 5 cohorts of 8 subjects each randomized 6:2 (S315:Placebo(0.9% Sodium Chloride)) with escalation of a fixed dose of S315
  Interventions: Drug: 0.9% Sodium Chloride (NaCl)

INTERVENTIONS:
Drug: S315 — Human monoclonal antibody against Diphtheria Toxin
  Arms: S315 human monoclonal antibody
Drug: 0.9% Sodium Chloride (NaCl) — Placebo 0.9% Sodium Chloride (NaCl)
  Arms: 0.9% sodium chloride (NaCl)

SUMMARY:
This study will examine the use of a single infusion of S315 at different doses in healthy volunteers to help understand its safety and tolerability. S315 is a monoclonal antibody that is being developed for treatment of diphtheria. The study will assess for any side effects when S315 and will also look at the levels of S315 in the blood over time.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent and able to effectively communicate with the Investigator and study personnel. A signed informed consent document (ICD) must be on file prior to initiating the screening procedures.

   Willing and able to complete all study requirements, restrictions, visits and procedures.
2. Age 18 to 55 years, inclusive.
3. Weight 50 kg to 90 kg, inclusive.
4. Systolic blood pressure less than 140 mmHg and diastolic less than 90 mmHg on two separate readings at least one minute apart.
5. Women of child bearing potential, defined as all women physiologically capable of becoming pregnant must agree not to become pregnant and must use a method of birth control during the entire study.

   Women of non-child bearing potential may be included. Women are considered post-menopausal and not of childbearing potential if, they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile or have had surgical total hysterectomy or tubal ligation at least six weeks ago.
6. Males of reproductive potential must use a barrier method of contraception during the course of the study.
7. Screening laboratory values must meet the following criteria:

   * White blood cell (WBC) 3.5 - Upper Limit of Normal (ULN)
   * Platelets > 100,000/mm3
   * Hemoglobin ≥ Lower Limit of Normal (LLN)
   * Creatinine ≤ ULN
   * Aspartate Aminotransferase (AST) ≤ ULN
   * Alanine Aminotransferase (ALT) ≤ ULN
   * Alkaline Phosphatase ≤ ULN
   * Bilirubin ≤ ULN
   * HgbA1c

Exclusion Criteria:

* 1. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.

  2. History of or any current medical condition that could compromise the safety of the participant in the study, as determined by the Investigator.

  3. History of suicidal behavior within 12 months prior to screening.

  4. Donated blood or plasma within 60 days prior to dosing.

  5. Clinically significant gastrointestinal, cardiovascular, neurologic, psychiatric, substance abuse, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease, as determined by the Investigator.

  6. Drug or alcohol abuse within previous 12 months or a positive test at screening and at Day -1 within 24 hours of study product administration.

  7. History of a previous severe allergic reaction with generalized urticaria, angioedema or anaphylaxis.

  8. Physical finding on examination considered clinically significant such as murmur (other than functional), hepatosplenomegaly, lymphadenopathy or focal neurological deficit.

  9. Urinalysis positive for > trace protein, > 5 Red Blood Cell (RBC)/hpf or > 5 WBC/hpf.

  10. Positive serology for HIV antibody, Hepatitis C Virus (HCV) antibody or Hepatitis B surface antigen at screening.

  11. Positive serum pregnancy test during screening or within 24 hours of study product administration, or an unwillingness to undergo pregnancy testing.

  12. Pregnant within 6 months or breast-feeding within 3 months prior to screening.

  13. Receipt of licensed vaccine containing diphtheria toxoid (Td, Tdap, pneumococcal conjugate vaccines, meningococcal conjugate vaccines) within the last year.

  14. Treatment with another investigational drug or other intervention within 30 days from screening.

  15. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the subject participating in the study.

  16. Safety laboratory abnormalities at Screening or Day -1, which are clinically significant as determined by the Investigator.

  17. Tobacco, e-cigarettes, and/or nicotine use within 30 days prior to screening confirmed by urine cotinine test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
The number of Participants with adverse events as assessed by the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table (Draft revised November 2007) adapted by the Division of Microbiology and Infectious Diseases, NIAID, NIH. | Day -1 through Day 60
  Adverse events assessed for safety

SECONDARY OUTCOMES:
Serial measurements of S315 concentration in the serum. | Day 1 pre-dose and Day 1, Day 2, Day 4, Day 8, Day 15, Day 22, day 29, Day 43 and Day 60 post-dose
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: John Z Sullivan-Bólyai, MD, MPH, Study Director — MassBiologics of the University of Massachusetts; Ronald Goldwater, MD, Principal Investigator — Parexel
Locations (1):
- Parexel Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith HL, Cheslock P, Leney M, Barton B, Molrine DC. Potency of a human monoclonal antibody to diphtheria toxin relative to equine diphtheria anti-toxin in a guinea pig intoxication model. Virulence. 2016 Aug 17;7(6):660-8. doi: 10.1080/21505594.2016.1171436. Epub 2016 Apr 12. PMID 27070129
- [Derived] Sullivan-Bolyai JZ, Allen LB, Cannon R, Cohane KP, Dunzo E, Goldwater R, StCyr K, Wang Y, Klempner MS. A Phase 1 Study in Healthy Subjects to Evaluate the Safety and Pharmacokinetics of a Human Monoclonal Antibody (S315) Against Diphtheria Toxin. J Infect Dis. 2025 Sep 15;232(3):534-539. doi: 10.1093/infdis/jiae499. PMID 39570031